CLINICAL TRIAL: NCT02529332
Title: Effect of Omega-3 Supplementation in Patients With Smell Dysfunction Following Endoscopic Pituitary Tumor Resection
Brief Title: Omega-3 Supplementation for Smell Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Zara M. Patel, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00076285
Record Dates: First submitted 2015-08-07; First posted 2015-08-20 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Sellar/Parasellar Tumor; Smell Dysfunction
Keywords: Endoscopic Sellar/Parasellar Tumor Resection
MeSH Terms: conditions — Olfaction Disorders | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 Supplementation Group (Experimental): Omega-3 supplementation
  Interventions: Dietary Supplement: Omega-3
- Control Group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Omega-3 — Nature Made Ultra Omega3 Fish Oil 1400mg softgels contains 1000mg of omega 3 per serving. Participants will be instructed to take twice daily for 6 months.
  Arms: Omega-3 Supplementation Group

SUMMARY:
Omega-3 supplementation has been shown to have neuroprotective and potentially anti-inflammatory properties in both central and peripheral nerve injuries. The investigators are studying to see if omega-3 supplementation will affect olfactory (smell) function in patients with olfactory dysfunction following endoscopic removal of pituitary tumors.

ELIGIBILITY:
Inclusion Criteria:

* sellar/parasellar tumor scheduled to undergo endoscopic transnasal transsphenoidal resection
* 18 years of age or older
* English speaking

Exclusion Criteria:

* Currently using blood thinning agents (aside from NSAIDs or cardioprotective ASA)
* elevated AST, ALT, or alk phos >10% outside of normal range, if randomized to omega-3 group
* diabetes, if randomized to omega-3 group and not already on omega-3 prescribed by another provider
* unable to provide informed consent due cognitive deficiencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Difference in Olfactory Function at baseline, based upon tumor type (i.e. functional vs. non-functional tumor) | Baseline (pre-tumor resection)
  The University of Pennsylvania Smell Identification Test (UPSIT) will be used to determine baseline olfactory function prior to sellar/parasellar tumor resection for all subjects.The test consists of a total of 40 "scratch and sniff" strips which the individual must select the correct odor from four choices. The test is scored out of 40 items. The number of correct answers regarding the smells being experienced is the subject's score. The higher the score the better the sense of smell.
Change in Olfactory Function over 6-month post-op period | Baseline (pre-tumor resection), at 6 months (post-tumor resection)
  The University of Pennsylvania Smell Identification Test (UPSIT) will be used to determine baseline olfactory function prior to sellar/parasellar tumor resection for all subjects.The test consists of a total of 40 "scratch and sniff" strips which the individual must select the correct odor from four choices. The test is scored out of 40 items. The number of correct answers regarding the smells being experienced is the subject's score. The higher the score the better the sense of smell. A change in UPSIT scores of 10% or greater indicates a clinically significant improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Zara M Patel, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Emory University Hospital, Atlanta, Georgia